CLINICAL TRIAL: NCT04709211
Title: A Comparative Study Between Postoperative Analgesia of Fascia Iliaca Compartment Block and Anterior Quadratus Lumborum Block in Proximal Femur Fracture
Brief Title: Fascia Iliaca Compartment Block Versus Anterior Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Assistant professor of Anaesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU M D 260/2020
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I: Facia Iliaca block (Active Comparator): patients will receive Ultrasound-guided Facia Iliaca Block using bupivacaine 0.25%
  Interventions: Procedure: Facia Iliaca block
- Group Q: Anterior Quadratus lumbroum block (Active Comparator): patients will receive Ultrasound-guided Anterior Quadratus Lumbroum block using bupivacaine 0.25%
  Interventions: Procedure: Anterior Quadratus Lumbroum block; Drug: bupivacaine

INTERVENTIONS:
Procedure: Facia Iliaca block — patients will receive Ultrasound-guided Facia Iliaca block using 50 ml 0f Bupivacaine 0.25%
  Arms: Group I: Facia Iliaca block
Procedure: Anterior Quadratus Lumbroum block — patients will receive Ultrasound-guided Anterior Quadratus Lumbroum block using 50 ml 0f Bupivacaine 0.25%
  Arms: Group Q: Anterior Quadratus lumbroum block
Drug: bupivacaine — bupivacaine
  Arms: Group Q: Anterior Quadratus lumbroum block

SUMMARY:
Fractures of the femur are common orthopaedic emergency especially in the geriatric population and central neuraxial blocks are the preferred technique for providing anaesthesia. However, limb immobility and extreme pain are the deterrents for ideal positioning for these procedures. postoperative pain is a nightmare so adequate analgesia has been advocated to reduce the pain. in this study, Facia Iliaca compartment block will be compared to anterior Quadratus lumborum block, both will be done Ultrasound-guided using Bupivacain0.25% for postoperative analgesia at the end of the surgery.

DETAILED DESCRIPTION:
In this prospective, randomized, comparative study patients will be equally divided into two equal groups; GroupI: patients will receive Ultrasound-guided Facia Iliaca compartment block with 50 ml 0.25%bupivacaine at the end of surgery Group Q: patients will receive Ultrasound-guided anterior Quadratus lumborum block with 50 ml 0.25%bupivacaine at the end of surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA II to IV
* Both sexes
* scheduled for fracture femur surgeries

Exclusion Criteria:

* patients with bleeding disorders and coagulopathy
* infection at the injection site
* known allergy to local anaesthetics
* patients with multiple fractures
* patients with pre-existing myopathy or neuropathy
* patients with significant cognitive dysfunction
* patients who receive long-acting opioids preoperatively

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
first request of analgesia | 48 hours postoperative
  the time the patient felt pain and asked for analgesics

SECONDARY OUTCOMES:
total opioid consumption | 48 hours postoperative
  total dose of fentanyl used

CONTACTS AND LOCATIONS:
Overall Officials: Fathy M Tash, MD, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No